CLINICAL TRIAL: NCT02074735
Title: Citicoline for Alcohol Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 072012-088
Record Dates: First submitted 2014-02-26; First posted 2014-02-28 (Estimated); Results first posted 2018-07-24 (Actual); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Alcohol Dependence
Keywords: alcohol dependence; alcohol abuse
MeSH Terms: conditions — Alcoholism | interventions — Sugars; Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo schedule will mimic the schedule of the active comparator citicoline. Placebo will be started at the randomization visit (week 0, mimicking 500 mg/day of citicoline), then increased at week 2 to mimic 1000 mg/day citicoline, then increased to mimic 1500 mg/day of citicoline at week 4, and then increased to mimic 2000 mg/day of citicoline at week 6 until the end of week 12.
  Interventions: Drug: Placebo
- Citicoline (Active Comparator): Citicoline will be started at 500 mg/day at the randomization visit (week 0), then increased to 1000 mg/day at week 2, then 1500 mg/day at week 4, and then 2000 mg/day at week 6 until the end of week 12.
  Interventions: Drug: Citicoline

INTERVENTIONS:
Drug: Placebo — Inactive ingredient matching the active comparator in appearance
  Other Names: Sugar pill
  Arms: Placebo
Drug: Citicoline — Citicoline is an over-the-counter nutritional supplement that is used for neuroprotective effects. It is a naturally occurring neurochemical in the human body.
  Other Names: CDP-choline; cytidine diphosphate-choline
  Arms: Citicoline

SUMMARY:
The purpose of this study is to determine if citicoline, as an add-on therapy, will help reduce alcohol use in outpatients with alcohol dependence.

DETAILED DESCRIPTION:
A total of 62 outpatients with alcohol dependence will be enrolled in a 12-week, randomized, placebo-controlled trial. Participants will be randomized to receive either placebo or citicoline.

Throughout the study, participants will be asked about their alcohol use and any withdrawal or craving symptoms. Depressive symptoms will be measured as well. Cognition and memory will be measured as well with a neurocognitive battery. Blood will be drawn at study start and week 12 to measure liver enzyme levels.

Appointments will be weekly for the entire study. Participants will have a physician follow-up at every study appointment.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-75 years old with diagnosis of alcohol dependence
* Average alcohol use of at least 28 drinks per week and at least 7 heavy drinking days (defined as 4 or more drinks/day for women, 5 or more drinks/day for men) in the past 28 days
* No alcohol use within 72 hours of randomization (maximum abstinence 7 days)
* CIWA-Ar (withdrawal scale) score less than or equal to 8 at randomization (consistent with minimal or no withdrawal symptoms and medication probably not needed)

Exclusion Criteria:

* Vulnerable populations including individuals with intellectual disability or dementia, prison or jail inmates, pregnant or nursing women, or women of childbearing age who will not use acceptable forms of birth control
* History of arrhythmias
* Myocardial infarction or coronary artery bypass graft surgery in the past 6 months
* Active angina or blood pressure >170/105
* High risk for suicide (defined as suicide attempt in past 6 months, or current suicidal ideation with plan and intent)
* High risk of violence toward others (defined as assault in past 6 months, or violent thoughts with evidence of plan and intent)
* Intensive outpatient treatment for substance abuse (AA, NA meetings or weekly therapy/counseling for substance use for at least 28 days prior to randomization will be allowed)
* Dependence (not just abuse) on substances other than alcohol or nicotine
* History of delirium tremens or other sever alcohol withdrawal symptoms, history of cirrhosis or AST or ALT >3 times normal, or other unstable medical condition (e.g. uncontrolled diabetes)
* History of bipolar disorder or schizophrenia
* Current major depressive episode (past episodes and current milder depressive symptoms allowed) or other psychiatric disorder that should be a major focus of treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherwood Brown, M.D., Ph.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The University of Texas Southwestern Medical CEnter, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Citicoline
Started | 29 | 33
Completed | 26 | 29
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Citicoline | Total
Number analyzed (Participants) | 29 | 33 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.79 (9.51) | 48.70 (8.92) | 46.87 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 24 | 25 | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 17 | 16 | 33
  Caucasian | 9 | 14 | 23
  Hispanic | 3 | 2 | 5
  Other | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 33 | 62

OUTCOME MEASURES:

1. Primary Outcome: Heavy Drinking Days Per Week
Description: Heavy drinking days are defined as "4 or more drinks for women, 5 or more drinks for men in a single day". Participants self-reported the type and amount of alcohol consumed during each assessment period. From this information, number of standard drinks per day was calculated using the following formula: "(number of drinks) x (oz per drink) x (alcohol by volume or ABV)". The average number of heavy drinking days was calculated by dividing the number of heavy drinking days per week by the number of days in the assessment period.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: days/week
Arm/Group | Placebo | Citicoline
Number analyzed (Participants) | 26 | 29
days/week | 0.23 (0.30) | 0.33 (0.38)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Placebo | Citicoline
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/29
Other Adverse Events (participants affected / at risk) | 15/26 | 22/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=26) | Citicoline (N=29)
Dry mouth (General disorders) | 1 | 4
Nausea (Gastrointestinal disorders) | 2 | 4
Headache (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 1
Drowsiness (Vascular disorders) | 4 | 5
Increased energy (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 3
Bruising (Injury, poisoning and procedural complications) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Fatigue (General disorders) | 1 | 0
Increased appetite (General disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Stomachache (Gastrointestinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No